CLINICAL TRIAL: NCT07387211
Title: Study SARS-CoV-2-CZ-PREVAL-II - Arm of the Olomouc Region Study to Quantify the Presence of Antibodies and Cellular Immunity Against SARS-CoV-2 in the Population of Persons Participating in the SARS-CoV-2-CZ-PREVAL Study in 2020
Brief Title: Study SARS-CoV-2-CZ-PREVAL-II - Arm of the Olomouc Region
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Collaborators: Palacky University (Other); University Hospital Olomouc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 34909
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: SARS-CoV-2; SARS-CoV-2 (COVID-19) Infection
Keywords: SARS-CoV-2
MeSH Terms: conditions — COVID-19; Infections | interventions — Blood Specimen Collection; Body Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants of the SARS-CoV-2-CZ-Preval study from the Olomouc region (Other): Population of persons involved in the SARS-CoV-2-CZ-Preval study in 2020 in the Olomouc region
  Interventions: Procedure: Blood sampling; Procedure: Gargle sampling; Other: Questionnaire completion; Diagnostic Test: Body temperature measurement

INTERVENTIONS:
Procedure: Blood sampling — Venous blood sampling three times on three visits of the study.
Procedure: Gargle sampling — Gargle sampling using GARGTEST sampling kit on three visits of the study and also gargle self-sampling using GARGTEST sampling kit at 14-day intervals between the study visits.
Other: Questionnaire completion — Patient will complete questionnaire on each visit on SARS-CoV-2 infections and vaccinations
Diagnostic Test: Body temperature measurement — Body temperature will be measured by healthcare professional at each visit to exclude patients with acute infection.

SUMMARY:
The aim of the study is to find the proportion of people in the population of the Olomouc Region with the presence of IgG (or IgM) antibodies against the S and N antigens of the SARS-CoV-2 virus, therefore people who have already encountered the SARS-CoV-2 virus with manifest antibody formation, or people who have undergone vaccination against COVID-19.

DETAILED DESCRIPTION:
Study has three study visits. First two visits are three months apart. Second and third visits are five months apart. On each study visit participant will provide venous blood sample and saliva sample obtained by gargling with the use of GARGTEST sampling kit. Participant will also fill in a questionnaire about SARS-CoV-2 infections and vaccinations. Site staff will measure the body temperature of the patient to exclude a patient with an acute infection. Blood sample will be used for the assessment of antibodies and cellular immunity of SARS-CoV-2. Part of the blood will be biobanked for the future SARS-CoV-2 biomarker determination. Gargling sample will be used for the demonstration of the pathogen on mucous membranes. Gargle self-sampling using GARGTEST sampling kit will be done by participants at 14-day intervals between the study visits. For gargle sample RT-PCR (real time polymerase chain reaction) will be done to determine the patogen presence.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the SARS-CoV-2-CZ-PREVAL study and venous blood examined as part of this study
* Signed study informed consent and consent to the processing of personal data
* Adults (age 18 and over)
* Willingness to complete the questionnaire

Exclusion Criteria:

• Participant with acute health problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2484 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

PRIMARY OUTCOMES:
The proportion of people in the population of the Olomouc Region with the presence of antibodies against the SARS-CoV-2 virus | 12 months
  The proportion of people in the population of the Olomouc Region with the presence of IgG (or IgM) antibodies against the S and N antigens of the SARS-CoV-2 virus, therefore people who have already encountered the SARS-CoV-2 virus with manifest antibody formation, or people who have undergone vaccination against COVID-19.

SECONDARY OUTCOMES:
Quantification of the level/presence of cellular immunity | 12 months
  Quantification of the level/presence of cellular immunity will be done from venous blood.
Verification of the presence of the SARS-CoV-2 virus | 12 months
  Verification of the presence of the SARS-CoV-2 virus on the mucous membranes of the oral cavity and pharynx using a PCR (polymerase chain reaction) test
Proportion of people with an asymptomatic course of SARS-CoV-2 disease | 12 months
  Proportion of people with an asymptomatic course of the disease - a combination of antibody tests, questionnaire surveys and data from the Institute of Health Information and Statistics of the Czech Republic will be used to assess this outcome.
Quantification of the presence of antibodies and the presence of cellular immunity | 12 months
  Quantification of the presence of antibodies and the presence of cellular immunity according to risk factors and time interval since infection/immunization

CONTACTS AND LOCATIONS:
Overall Officials: Marian Hajduch, MD, PhD, Study Director — Palacky University Olomouc
Locations (1):
- University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No